CLINICAL TRIAL: NCT00610532
Title: Evaluating Transporter Protein Inhibitors in Patients With Epilepsy
Brief Title: Evaluating the Transporter Protein Inhibitor Probenecid In Patients With Epilepsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigators decided not to continue
Sponsor: Jim McAuley (Other)
Responsible Party: Sponsor-Investigator, Jim McAuley, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2005H0170
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Epilepsy
Keywords: pharmacoresistance; healthy volunteers
MeSH Terms: conditions — Epilepsy | interventions — Phenytoin; Probenecid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): intravenous phenytoin alone
  Interventions: Drug: phenytoin
- B (Experimental): intravenous phenytoin plus probenecid
  Interventions: Drug: phenytoin and probenecid

INTERVENTIONS:
Drug: phenytoin — intravenous phenytoin (15 mg/kg) single dose
  Arms: A
Drug: phenytoin and probenecid — intravenous phenytoin (15 mg/kg) single dose and oral probenecid 2000 mg single dose
  Arms: B

SUMMARY:
The study is being done to understand why some patients with epilepsy (disease of recurrence of seizures) do not respond very well to drug treatment with anticonvulsants.

Despite the availability of many anticonvulsants, about 30% of patients with epilepsy are resistant to them. The cause of the resistance is not clear, but one of the reasons could be an increased amount of proteins in the cells of the body called transporter proteins.

Transporter proteins are a group of proteins that help to defend the body against toxins, including drugs, by pumping them out of the cells. Studies have shown that the number of transporter proteins is higher in the parts of the brain that trigger seizures when compared to other parts of the brain.

Studies in animals have shown that taking an anticonvulsant with an inhibitor (meaning "to stop" or "to reduce") of a transporter protein can increase the concentration of that anticonvulsant inside the brain cells. The main purpose of the study is to determine if taking an anticonvulsant and a transporter protein inhibitor will change the brain concentration of the anticonvulsant.

In this study, a single dose of phenytoin (Dilantin® is a brand name anticonvulsant which has phenytoin as its active ingredient), a commonly used anticonvulsant, will be given once by itself, and then will be given a separate time with a single (i.e. one time only) dose of probenecid. Probenecid, a medicine used commonly to treat gout (a disease of increased uric acid), is known to be an inhibitor of transporter proteins. The study will use electroencephalogram or EEG (recording of brain wave activities) to determine if the EEG pattern when probenecid is given, will be different from the EEG pattern when phenytoin is given alone. This will suggest that probenecid has affected the brain concentration of phenytoin.

DETAILED DESCRIPTION:
About 30% of patients with epilepsy are refractory to medical treatment (pharmacoresistant epilepsy). The cause of which is multifactorial. Multidrug resistance (MDR) causes decreased uptake of medicines in tissues. MDR occurs because of overexpression of a family of transporter proteins that act as a physiological defense mechanism that pumps toxins out of cells. Two groups of transporters, P-glycoprotein (PGP) and multidrug resistance-associated proteins (MRP), are important gatekeepers in the blood brain barrier. PGP and MRP are overexpressed in the brain tissue of pharmacoresistant patients with partial epilepsy and many antiepileptic drugs (AEDs) are substrates for PGP, MRP or both.

It is logical to try to apply these observations to clinical practice. We hope that through co-administration of an inhibitor of transporter proteins, we can increase the CNS concentrations of AEDs, and subsequently improve seizure control. However, before this, it is critical to demonstrate that a transporter protein inhibitor can increase the concentration of AEDs in human brain.

Probenecid is an MRP inhibitor while phenytoin is an MRP substrate. Evaluating whether probenecid can increase the CNS concentration of PHT can potentially be achieved noninvasively by using pharmaco-EEG.

We plan to estimate the effect of probenecid (a transporter protein inhibitor) on the quantitative EEG recordings when it is administered to patients with pharmacoresistant epilepsy and in normal healthy volunteers.

We plan to recruit two groups of 10 subjects each, normal volunteers and patients with pharmacoresistant epilepsy. They will undergo two treatment regimens; EEG recording after administration of intravenous phenytoin only and again after pre-dosing them with probenecid.

ELIGIBILITY:
Inclusion Criteria:

* Men with pharmacoresistant partial epilepsy defined as failure of two or more AEDs at a reasonable therapeutic dose
* Patient is able to understand and sign a consent form and able to keep a seizure calendar
* Patient is older than 18 years of age
* Patient is otherwise healthy by laboratory and physical examination

Exclusion Criteria:

* Patient is currently taking phenytoin
* Patient has a history of an adverse reaction to phenytoin
* Patient has a history of gout disease, peptic ulcer disease, blood dyscrasias, or uric acid kidney stones
* Patient has an allergy to sulfa drugs or probenecid
* Patient has been exposed to probenecid or another known transporter inhibitor (verapamil, progesterone, etc) in the three months prior to enrollment
* Patient has a history of renal impairment (creatinine clearance < 50 ml/min)
* Patient has a history of diabetes and is taking oral sulfonylurea agents

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W McAuley, PhD, Principal Investigator — Ohio State University; Bassel F Shneker, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between Feb 2006 and Sept 2007.
Groups:
- All Study Participants: All study participants progressed from receiving intravenous phenytoin alone to intravenous phenytoin plus probenecid.
Period: Intravenous Phenytoin Alone
Arm/Group | All Study Participants
Started | 8
Completed | 8
Not Completed | 0
Period: Intravenous Phenytoin Plus Probenecid
Arm/Group | All Study Participants
Started | 7 (one participant dropped out between periods)
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants progressed from intravenous phenytoin alone to intravenous phenytoin plus probenecid
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Quantitative EEG Recordings
Time Frame: end of each treatment
Population: No data was analyzed because the study was terminated by the investigators after they decided not to continue the project
Groups:
- Intravenous Phenytoin Alone: intravenous phenytoin alone
- Intravenous Phenytoin Plus Probenecid: intravenous phenytoin plus probenecid
Arm/Group | Intravenous Phenytoin Alone | Intravenous Phenytoin Plus Probenecid
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Phenytoin Alone | Intravenous Phenytoin Plus Probenecid
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
problems with measurement led to uninterpretable data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No